CLINICAL TRIAL: NCT04112979
Title: Effects of Intraoperative Auditory Stimulation on Pain and Agitation at Awakening After Pediatric Adenotonsillectomy - 4 Arms, Double-blinded, Randomized, Controlled Clinical Trial
Brief Title: Auditory Intraoperative Stimulation Effects on Pain and Agitation at Awakening (AUDIOPAW)
Acronym: AUDIOPAW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Burlo Garofolo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC 36/18
Record Dates: First submitted 2019-08-06; First posted 2019-10-02 (Actual); Last update posted 2019-10-02 (Actual); Status verified 2019-10

CONDITIONS: Procedural Anxiety; Procedural Pain; Adenotonsillitis
Keywords: Auditory stimulation; adenotonsillectomy; pain; agitation; awakening
MeSH Terms: conditions — Pain, Procedural; Pain; Psychomotor Agitation | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Auditory stimulation 1 (Music) (Experimental): 45 deciBel Sensation Level (dB SL), normalized, high-frequency sampled W.A. Mozart Symphony n°4 in D K19 and n°5 in B-flat K22 (from Mozart Symphonies Vol. I - Adam Fisher, Dacapo Records, Frederiksberg C., Denmark, 2013)
  Interventions: Behavioral: Music
- Auditory stimulation 2 (Mother's lap) (Experimental): 45 dB SL, normalized and filtered, high-frequency sampled heartbeat sound, 75 bpm tempo, looped
  Interventions: Behavioral: Mother's lap
- Soundproof earplugs (Experimental): Disposable foam earplugs with a noise attenuation of at least 30 deciBel (dB)
  Interventions: Behavioral: Soundproof earplugs
- No stimulation (No Intervention): Current standard of care

INTERVENTIONS:
Behavioral: Music — 45 dB SL, normalized, high-frequency sampled W.A. Mozart Symphony n°4 in D K19 and n°5 in B-flat K22 (from Mozart Symphonies Vol. I - Adam Fisher, Dacapo Records, Frederiksberg C., Denmark, 2013)
  Arms: Auditory stimulation 1 (Music)
Behavioral: Mother's lap — 45 dB SL, normalized and filtered, high-frequency sampled heartbeat sound, 75 bpm tempo, looped
  Arms: Auditory stimulation 2 (Mother's lap)
Behavioral: Soundproof earplugs — Disposable foam earplugs with a noise attenuation of at least 30 dB
  Arms: Soundproof earplugs

SUMMARY:
Adenotonsillectomy (AT) is one of the most common pediatric surgical procedures. The management of postoperative pain and agitation after AT is still a controversial issue. Safety considerations limit the use of opioids and non-steroidal anti-inflammatory drugs, leading to inadequate control of the high levels of postoperative pain experienced by AT patients. Along with pain killers, non-pharmacological strategies have remarkable impact on pain management in children. A systematic review and meta-analysis published in The Lancet in 2015 on adult patients suggest that auditory stimulation with music in the perioperative setting, and even when patients are under general anaesthesia, can reduce postoperative pain, anxiety, and analgesia needs. The authors concluded that there is sufficient evidence to implement auditory stimulation in the treatment of all adult surgical patients, regardless of the mode of administration. Up to now, no research has investigated the effects of intraoperative auditory stimulation on pain and agitation upon awakening after AT in the pediatric population. Objective of this study is to determine the effects of intraoperative auditory stimulation on pain and agitation upon awakening after pediatric AT.

ELIGIBILITY:
Inclusion criteria:

* age 2 to 17 years old
* scheduled for adenotonsillectomy
* recent audiometry and tympanometry evaluation (<1 month)

Exclusion Criteria:

* no informed consent
* other combined surgical procedures
* comorbidities (e.g. congenital anomalies of the head-and-neck, psychomotor delay, autism spectrum disorders)
* American Society of Anesthesiologists (ASA) Classification score >2
* ongoing chronic pharmacological therapy
* first language not Italian
* environmental noise exceeding limits in the operating room

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 115 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-24 (Actual)

PRIMARY OUTCOMES:
Pain score (Wong-Baker Faces Pain Rating Scale), self-administered (collaborative children between 3 and 8 years) | Within 10 minutes after awakening
  Pain score for collaborative children between 3 and 8 years will be evaluated with the self-administered Wong-Baker Faces Pain Rating scale, ranged 0-10.
  Higher scores correspond to higher levels of pain.
Pain score (Visual Analogue Scale), self-administered (collaborative children >=8 years) or administered by parents (non-collaborative children >=8 years) | Within 10 minutes after awakening
  Pain score for >=8 years old children will be evaluated with Visual Analogue Scale (self administered if collaborative; administered by parents if non-collaborative children), ranged 0-10.
  Higher scores correspond to higher levels of pain.
  In accordance with previous studies (Ferreira-Valente et al. Validity of four pain intensity rating scales. Pain 2011;152:2399-2404), the scores of Wong-Baker Faces Pain Rating scale and Visual Analogue Scale will be considered comparable and combined in one outcome variable.
Pain score (Face, Legs, Activity, Cry, Consolability scale), evaluated by parents (for children <=3 years) | Within 10 minutes after awakening
  For children <=3 years, pain score will be evaluated by parents using the Face, Legs, Activity, Cry, Consolability (FLACC) scale, ranged 0-10.
  Higher scores correspond to higher levels of pain.
Pain score (Children's Hospital of Eastern Ontario Pain scale), evaluated by parents (for non-collaborative children between 3 and 7 years) | Within 10 minutes after awakening
  For non-collaborative children between 3 and 7 years, pain score will be evaluated by parents using the Children's Hospital of Eastern Ontario Pain (CHEOPS) scale, ranged 0-10.
  Higher scores correspond to higher levels of pain.
  In accordance with previous studies, the scores of the Face, Legs, Activity, Cry, Consolability (FLACC) scale and of the Children's Hospital of Eastern Ontario Pain (CHEOPS) scale will be considered comparable and combined in one outcome variable.

SECONDARY OUTCOMES:
Agitation | Within 10 minutes after awakening
  Evaluated using the Paediatric Anesthesia Emergence Delirium (PAED) scale, ranging form 0 to 20. Higher scores correspond to higher levels of agitation.
Frequency of use of pain killer drugs | Within 6 hours after the awakening
  Number of postoperative pain killers drugs administered

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Muzzi, MD, Study Chair — IRCCS Burlo Garofolo
Locations (1):
- Institute for Maternal and Child Health - IRCCS Burlo Garofolo-, Trieste, Italy

REFERENCES:
- [Derived] Muzzi E, Ronfani L, Bossini B, Lezcano C, Orzan E, Barbi E. Effects of Intraoperative Auditory Stimulation on Pain and Agitation on Awakening After Pediatric Adenotonsillectomy: A Randomized Clinical Trial. JAMA Otolaryngol Head Neck Surg. 2021 Jul 1;147(7):638-645. doi: 10.1001/jamaoto.2021.0870. PMID 34014258